CLINICAL TRIAL: NCT06339736
Title: Treatment Outcomes in Patients With Muscular Temporo-mandibular Joint Disorders
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Rossana Izzetti, Researcher at the Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine of the University of Pisa, Principal Investigator, University of Pisa
Other Study IDs: 23815
Record Dates: First submitted 2024-03-21; First posted 2024-04-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: TMD; TMD/Orofacial Pain
Keywords: Temporomandibular Joint Disorders; Quality of Life; Oral Health; Oral Health-Related Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- M-TMD group: Patients with a diagnosis of muscular TMDs performed according to DC/TMD criteria
  Interventions: Other: Questionnaires administered to all study participants
- CTRL group: A control group of subjects with a negative history for TMDs
  Interventions: Other: Questionnaires administered to all study participants

INTERVENTIONS:
Other: Questionnaires administered to all study participants — Ten treatment sessions were performed, which initially involved muscular stretching and relaxation exercises and then strengthening and endurance exercises to achieve stabilization. An oral splint was applied to he upper dental arch.

SUMMARY:
The aim of the present study was to assess the treatment outcomes in patients affected by M-TMDs in terms of pain scores assessed with pressure pain threshold (PPT). The levels of de-pression, anxiety and the Oral-Health Impact profile were also assessed and compared to healthy controls. Patients with a clinical diagnosis of M-TMDs and a control group of healthy subjects were enrolled. At baseline, OHIP-14, PHQ-9 and GAD-7 were administered. PPT was registered at the level of masseter and temporalis muscles. The patients were then treated with oral splints and physio-kinesiotherapy following a standardized treatment protocol. At 6-months follow-up, PPT was registered, and the questionnaires were re-administered to compare treatment outcomes.

DETAILED DESCRIPTION:
Consecutive patients referred to the Unit of Dentistry and Oral Surgery for suspected TMD between January 2022 and December 2022 were enrolled. All the study participants signed an informed consent form to be included in the study.

Two study groups were identified:

* M-TMD group, including patients with a diagnosis of muscular TMDs;
* A control group of subjects with a negative history for TMDs. The inclusion criteria for patients in the M-TMD group were i) males or females >18 years, ii) systemically healthy patients, iii) clinical examination revealing a diagnosis of muscular TMD and/or positive history of muscular TMD, iv) patients willing to give informed consent, and v) compliance to the study follow-up. Patients with i) articular TMDs, ii) chronic diseases, iii) any psychiatric diagnosis under medication, iv) pregnant or lactating, and v) not willing to comply with the study protocol were excluded.

The subjects included in the control group were enrolled among the patients referred to the Unit of Oral Surgery of the Unit of Dentistry and Oral Surgery. The patients in the control group were i) males or females of age > 18 years, ii) systemically healthy patients, iii) clinical examination negative for pain in the masticatory muscles and negative for history of TMDs, and iv) patients willing to give informed consent and to be administered the study questionnaires.

After diagnosis confirmation of M-TMD according to the DC/TMD criteria, the patients were treated with the application of an oral splint on the upper dental arch associated with physio-kinesiotherapy.

The patients were administered OHIP-14, PHQ-9, and GAD-7 questionnaires to compare scores in the M-TMD patients versus healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* males or females >18 years of age
* systemically healthy patients
* clinical examination revealing a diagnosis of muscular temporo-mandibular joint disorder (TMD) and/or positive history of muscular TMD
* patients willing to give informed consent, and v) compliance to the study follow-up.

Exclusion Criteria:

* articular TMDs
* chronic diseases
* any psychiatric diagnosis under medication
* pregnant or lactating females
* not willing to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the Unit of Dentistry and Oral Surgery for suspected TMD
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of muscular pain on oral health | 6 months
  Assessment of Oral Health Impact Profile -14 (OHIP-14) questionnaire scores following treatment. Scores range between 0 (absence of oral health impairment) and 56 (severe oral health impact)
Evaluation of the impact of muscular pain on anxiety | 6 months
  Assessment of General Anxiety Disorder-7 (GAD-7) questionnaire scores following treatment. Scores range from 0 to 21. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety.
Evaluation of the impact of muscular pain on depression | 6 months
  Assessment of Patient Health Questionnaire-9 (PHQ-9) questionnaire scores following treatment. score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression)

SECONDARY OUTCOMES:
Changes in muscular pain | 6 months
  Changes in muscular pain following treatment assessed through pressure pain threshold

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided